CLINICAL TRIAL: NCT01658605
Title: A Phase II, 20-week, Multi-centre, Randomised, Double-blind, Placebo-controlled, Parallel Group Proof of Concept Study to Investigate the Efficacy and Safety of GSK1605786 for Treatment of Patients With Active Ulcerative Colitis
Brief Title: A Study to Investigate the Efficacy and Safety of GSK1605786 for Treatment of Patients With Active Ulcerative Colitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study CCX115383 has been terminated prior to enrolment of any patients. A decision was made by GSK to delay pursuit of this indication as the biology evolves.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 115393
Record Dates: First submitted 2012-05-24; First posted 2012-08-07 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Colitis, Ulcerative
Keywords: GSK1605786; ulcerative colitis; CCR9 antagonist; proof of concept
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- GSK1605786 (Experimental): Administered orally for 16 weeks in a 2:1 ratio
  Interventions: Other: Placebo
- Placebo (Placebo Comparator): Administered orally for 16 weeks in a 2:1 ratio
  Interventions: Drug: GSK1605786

INTERVENTIONS:
Drug: GSK1605786 — 500 mg twice daily administered orally
  Arms: Placebo
Other: Placebo — 500 mg twice daily administered orally
  Arms: GSK1605786

SUMMARY:
GSK1605786 is an oral antagonist specific for the chemokine receptor CCR9 in development for treatment of small bowel and colonic Crohn's disease (CD). The purpose of this Phase II proof of concept study is to investigate the efficacy and safety of GSK1605786 (500 mg twice daily) administered orally for 16 weeks for the treatment of patients with active ulcerative colitis (UC). A key secondary objective is to understand the mechanism by which GSK1605786 is acting and to this end samples will be collected to confirm the degree of inhibition of CCR9 on T lymphocytes in the blood of patients, and to explore the relationship between concentration of drug and changes in lymphocyte and antigen presenting cell populations in the peripheral circulation and in the colon. Patients recruited at specified investigational sites will be invited to participate in an optional sub-study to explore the effects of GSK1605786 on trafficking of technetium labelled T cells using Single Photon Emission Computerized Tomography (SPECT). Specifically, the technique will be used to follow trafficking to large intestine and thymus and findings linked to pharmacokinetics of GSK1605786, receptor occupancy and clinical efficacy outcomes

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 and over at the time of signing the informed consent.
* A female subject of child-bearing potential is eligible to participate if she agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until completion of the follow-up visit.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form, prior to any of the screening procedures including discontinuation of prohibited medication.
* At screening (visit 1): patients with a clinical history and examination suggestive of active UC for at least 3 months despite at least 2 weeks treatment with oral >2.4g/day mesalazine / mesalamine or equivalent.
* At screening/randomization (visit 2):

  * Presence of active UC spread beyond the rectum (inflammation extending ≥ 15cm from anal verge) as evidenced by flexible sigmoidoscopy or colonoscopy during the screening window.
  * AND MAYO score of 5 - 10 inclusive.
* AST and ALT < 2xULN; alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN

Exclusion Criteria:

* If female, is pregnant, has a positive pregnancy test or is breast-feeding.
* Confirmed diagnosis of celiac disease, those who follow a gluten-free diet to manage symptoms of suspected celiac disease and subjects with positive serologic test for Tissue transglutaminase, tTG.
* Subjects who have received immunisation with a live vaccine e.g. measles, mumps, rubella (each as in MMR vaccine), oral polio, varicella, yellow fever, within 4 weeks of screening and throughout the study, with the exception of influenza vaccine.
* Known or suspicion of CD, indeterminate colitis, microscopic colitis, ischaemic colitis or radiation-induced colitis, based on medical history, endoscopy and/or histological findings.
* Subjects with imminent need for surgery for UC in the opinion of the investigator.
* Subjects where assessment of MAYO score is likely to be confounded by previous surgery (for example colectomy, ileostomies, colostomies or rectal pouches).
* Subjects requiring enteral or parenteral feeding.
* Use of prohibited medications within their specified timeframes (see Section 9).

  * 5-Aminosalicylic acid enema: within 2 weeks of screening and throughout study
  * Topical (suppository) 5-Aminosalicylic acid: at screening and throughout study
  * Biologic use: within 12 weeks of screening and throughout study
  * Corticosteroids use: Oral, rectal or parenteral corticosteroids within 4 weeks of screening and throughout study
  * Antibiotics: Intravenous antibiotics within 8 weeks of screening and throughout study (oral antibiotics are permitted where they have been used for >4 weeks with stable dose for ≥2 weeks prior to screening)
  * Probiotics: within 4 weeks of screening (patients who initiated probiotics or prebiotics more than 4 weeks prior to screening should continue use throughout study)
  * NSAIDs: Within 7 days of screening and throughout the study (except low dose aspirin (≤325 mg/day) which may be continued for cardioprotection)
  * Digoxin: or related cardiac glycoside (e.g. digitoxin, deslanoside, lanatoside C, metildigoxin) use at any time during screening and throughout the study.
* Known HIV infection
* A positive HBsAg, Anti-HBc, or Hepatitis C antibody result at screening or documented positive result within 3 months of screening.
* Known varicella, herpes zoster, or other severe viral infection within 6 weeks of screening.
* Active or latent tuberculosis (TB) infection:

  * The subject has a history of TB disease or latent TB infection, in the absence of documented adequate therapy for same.
  * Suspicion of current TB disease (including extra pulmonary TB disease such as tuberculosis enteritis) or latent tuberculosis infection, as evidenced by positive QuantiFERON-TB Gold test, or T-SPOT.TB test.
* Current or chronic history of liver disease or known hepatic or biliary abnormalities including primary sclerosing cholangitis (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QTc ≥450 msec (≥480msec for those with Bundle Branch Block).

  * either QTcb or QTcf, machine or manual overread, males or females. The QT correction formula used to determine exclusion and discontinuation should be the same throughout the study.
  * based on single QTc value of ECG obtained over a brief recording period.
* The subject has a concurrent illness or disability that may affect the interpretation of clinical data, or otherwise contraindicates participation in this clinical study (e.g., an unstable cardiovascular, autoimmune, congenital or acquired immunodeficiency, renal, hepatic, pulmonary, endocrine, metabolic, gastrointestinal, haematologic, or neurological condition or mental impairment).
* The subject has current evidence of, or has been treated for a malignancy within the past 5 years (other than localised basal cell, squamous cell skin cancer, cervical dysplasia, or cancer in situ that has been resected).
* Use of any investigational drug within 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer) prior to screening
* Medical history of sensitivity to any of the components of GSK1605786 (microcrystalline cellulose, colloidal silicon dioxide, crospovidone, magnesium stearate, gelatin).
* Prior exposure to GSK1605786: Any previous exposure to GSK1605786 (formerly ChemoCentryx compound CCX282-B).
* Known positive stool culture for enteric pathogens
* Positive immunoassay for C. difficile.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period (with the exception of subjects involved in the optional scintigraphy sub-study, where no more than 700 mL of blood will be collected over the duration of the study, including any extra assessments that may be required).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2013-02 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of GSK1605786 at week 12 following twice daily administration at 500 mg in patients with active UC. | 12 weeks
  Ordinal response (remission, response, or no response) to treatment as assessed by the MAYO score at week 12.

SECONDARY OUTCOMES:
safety and tolerability of GSK1605786 in patients with active UC following repeat dosing continued for up to 16 weeks | 16 weeks
  Adverse events (AEs), Treatment effects on blood pressure, heart rate, electrocardiography (ECG) parameters and haematology, clinical chemistry and urinalysis findings
The time course of the efficacy of GSK1605786 | 16 Weeks
  Incidence of remission (MAYO score ≤ 2 with no individual subscale exceeding 1) at Week 12, incidence of response (MAYO score decreased for ≥ 3 points in comparison with baseline) at Week 12, change in partial MAYO score compared to baseline through week 16, change in SCCAI score compared to baseline through week 16, incidence of endoscopic remission (mucosal healing) rate at Week 12 (defined as proportion of patients with endoscopy score of 0 or 1 on the MAYO endoscopic sub-scale) and time to withdrawal and/or use of rescue medication
The anti-inflammatory activity of GSK1605786 in patients with active UC | 16 Weeks
  Circulating soluble biomarkers (CRP, CXL10), faecal calprotectin levels, receptor occupancy (CCR9 internalization).
The effects of GSK1605786 on quality of life in patients with UC | Baseline, week 12, week 16
  Quality of Life (IBDQ) Questionnaire.
The systemic pharmacokinetics (PK) of GSK1605786 following twice daily administration at 500 mg in patients with active UC. | DaysBaseline, week 4, week 8, week 12, week 16
  The maximum observed concentration (Cmax) on Day 28; Trough concentration (Cτ) on Day 28; Plasma clearance and volume of distribution estimated based on population pharmacokinetic analysis of healthy volunteers (historical data) and patient data, if possible
CCR9 occupancy (RO) in peripheral blood | 12 Weeks
  TECK/CCL25 and CCR9 expression in colon biopsy at baseline and at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- GSK Investigational Site, Leuven, Belgium
- GSK Investigational Site, Amsterdam, Netherlands
- United Kingdom (3):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, Southampton, Hampshire
  - GSK Investigational Site, Oxford, Oxfordshire